CLINICAL TRIAL: NCT05155423
Title: A Prospective Study of Performing MRI Simulation in Treatment Position in Spinal Stereotactic Body Radiation Therapy
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Elekta Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: PA18-0190; NCI-2021-11703 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2021-11-30; First posted 2021-12-13 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Spinal Metastases
MeSH Terms: interventions — Masks; Immobilization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: patient using mask for immobilization
  Interventions: Other: mask for immobilization
- group 2: patients using Elekta BodyFix
  Interventions: Other: Elekta BodyFix

INTERVENTIONS:
Other: mask for immobilization — mask for immobilization
  Groups: group 1
Other: Elekta BodyFix — Elekta BodyFix
  Groups: group 2

SUMMARY:
To learn the usefulness of performing MRI scans in different positions and learn the best practice for spinal stereotactic body radiation therapy (spinal SBRT) planning and dose delivery.

DETAILED DESCRIPTION:
1. Objectives

1. Assess the feasibility of performing MRI scans in the treatment position for accurate treatment planning and dose delivery in spinal stereotactic body radiation therapy (spinal SBRT).
2. Characterize the improved accuracy of image fusion between MRI and CT and its dosimetric impact when performing MRI scans in treatment position in spinal SBRT.
3. Assess the ability of MRI simulation to accurately target extended spinal targets beyond the current targeting limitations (>3 consecutive vertebral body levels)
4. Optimize the workflow of using MRI simulation in treatment planning and dose delivery.

ELIGIBILITY:
3.1. Inclusion Criteria

1. Greater than or equal to 18 years of age
2. Pathologically confirmed diagnosis of cancer, including, but not limited to non-small cell lung cancer, breast, prostate, renal cell, melanoma, gastrointestinal, sarcoma, thyroid, head and neck primary, and carcinoma of unknown primary
3. Signed informed consent
4. Willing to undergo 2 MRI simulations in one or multiple sessions, one with immobilization device, and the other without.
5. Patients undergoing spinal SBRT 3.2. Exclusion Criteria

a. Patient with a relative or absolute contraindication to MRI (such as pacemaker, etc.) b. Patients with significant instrumentation or cement at the site of interest causing artifact c. Inability to tolerate with immobilization device for greater than 30 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MDACC Cancer Participants
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2018-04-21 (Actual); Primary Completion 2026-05-24 (Estimated); Study Completion 2026-05-24 (Estimated)

PRIMARY OUTCOMES:
Performing MRI scans in the treatment position for accurate treatment planning. | through study completion, an average of 1 year
Performing MRI scans in the treatment position for dose delivery in spinal stereotactic body radiation therapy (spinal SBRT). | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Amol Ghia, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org